CLINICAL TRIAL: NCT01693081
Title: A Clinic-Based, Phase IIa, Double-Blind, Placebo- Controlled, Ascending-Dose, Multicentre Study of Safety, Tolerability, Efficacy and Pharmacokinetics of VR040 in Parkinson's Disease
Brief Title: Phase IIa Multicentre Study Investigating of VR040 in Parkinson's Disease
Acronym: VR040/2/003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Collaborators: Vectura Limited (Industry)
Responsible Party: Principal Investigator, Dr Donald Grosset, Consultant Neurologist, South Glasgow University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VR040/2/003
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; inhaled apomorphine; convert "off" to "on"
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VR040/Aspirair® inhaler (Active Comparator): VR040 was administered as an inhaled dry powder, in a dosage of 1.5, 2.3, 3.0 and 4.0mg, single dose given at each dose level.
  Interventions: Drug: VR040/Aspirair® inhaler
- Placebo (Placebo Comparator): Placebo was administered as an inhaled dry powder, matching to active comparator at dosages of 1.5, 2.3, 3.0 and 4.0mg, single dose given at each dose level.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: VR040/Aspirair® inhaler — Dry Powder inhaled apomorphine
  Other Names: Inhaled apomorphine
  Arms: VR040/Aspirair® inhaler
Drug: placebo
  Arms: Placebo

SUMMARY:
'Off periods' where people with Parkinson's disease are slow, stiff and unable to function are disabling, and a treatment which can converts people to a "on", good, able to function state would be extremely useful. We assessed safety, tolerability and efficacy of inhaled dry powder apomorphine (VR040) in a clinic-based study in this setting.

DETAILED DESCRIPTION:
Background: 'Off' periods increase as Parkinson's disease progresses and the benefits of standard therapy wane. Subcutaneous apomorphine rescues 'off' periods, but patient self-injection and adverse cutaneous effects are sometimes problematic.

Methods: We assessed safety, tolerability and efficacy of inhaled dry powder apomorphine (VR040) in a clinic-based Phase II study. Of 48 patients recruited at 9 sites, 47 were randomized 2:1 inhaled apomorphine:placebo. Respirable doses (drug predicted to reach the lung) ascending through 1.5mg, 2.3mg, 3.0mg, and 4.0mg until efficacy was achieved, were administered to patients in a practically defined 'off' state. The primary endpoint was the response in unified Parkinson's disease rating scale Part 3 (UPDRS 3), at the highest dose received by the patient. Secondary endpoints included time to 'on', the proportion of patients converting from 'off' to 'on', and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 30 and 90 years old with idiopathic PD for at least 5 years.
2. Voluntary written informed consent provided.
3. Willing and able to comply with study procedures.
4. Fulfilled steps 1 and 2 of the UK Brain Bank Criteria.
5. Classified as Hoehn and Yahr Stage II to IV in "on" state.
6. Motor fluctuations with recognisable "off" periods in control of motor symptoms, as assessed by the Motor Fluctuation Questionnaire.
7. Optimised oral therapy.
8. Dopaminergic responsiveness as defined by ≥ 30% improvement(reduction) in UPDRS III score compared with pre-dose value.

Exclusion Criteria:

1. Participated in a trial with an investigational product within prior 3 months.
2. Serious uncontrolled disease including serious psychological disorders.
3. Previous intolerance to apomorphine.
4. Previous significant complication from oral dopamine agonist therapy
5. Women lactating, pregnant or of child-bearing potential not using a reliable contraceptive method (eg, barrier, intrauterine device, abstinence).
6. Known HIV or active chronic hepatitis B or C infection.
7. Any clinically significant abnormality following review of screening observations
8. Patients who, in the Investigator's opinion, were unsuitable for the study for any reason.
9. Major ECG abnormalities.
10. Patients with a FEV1 ≤ 65% predicted.
11. Patients showing a postural decrease in systolic blood pressure (BP) of ≥20 mm Hg or showing significant clinical symptoms associated with orthostatic hypotension.
12. Patients with persistent arterial hypotension, with average systolic readings of ≤110 mm Hg.
13. Patients with persistent elevation of BP, with average systolic readings of ≥160 mm Hg.

    or average diastolic readings of ≥100 mm Hg.
14. Patients taking apomorphine at any time during these study visits, anabolic steroids,traditional antipsychotics (unless low dose) and vasodilators other than for the treatment of hypertension. The following atypical antipsychotics were permitted: Quetiapine (up to and including 50 mg per day), risperidone (up to and including 1 mg per day) and olanzapine (up to and including 2.5 mg per day).
15. Patients taking agents of the 5HT3 antagonist class including ondansetron, granisetron,dolasetron, palonosetron and alosetron.
16. Patients with existing cancer and those in remission for less than 5 years.
17. Patients with evidence (as ascertained from examination, tests or history) to indicate cardiovascular, gastrointestinal tract, liver, kidney, central nervous system, pulmonary system or bone marrow disorders that in the Investigator's opinion compromised patient safety.
18. Patients who were known non-responders to apomorphine treatment for "off" episodes(eg, in previous challenge tests or trials).
19. Patients with a history of drug or alcohol abuse in the 12 months prior to entry.
20. Patients with a history of clinically significant allergies to VR040 formulation constituents (including lactose and opioids) and domperidone.
21. Patients with signs or symptoms suggestive of psychosis, dementia, "Parkinson-plus" syndromes or unstable systemic disease.
22. Patients with history of stroke, seizure or other neurological conditions.
23. Patients with dyskinesia rated 4 in Item 32 of UPDRS IV assessment at Screening(dyskinesia present ≥76% of a waking day).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-03; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The maximum UPDRS 3 improvement from pre-dose to post-dose | 90 minutes
  The primary efficacy endpoint was the maximum UPDRS 3 improvement from pre-dose to post-dose at the highest dose used.

SECONDARY OUTCOMES:
Time to improvement from 'off' to 'on' | 90 minutes
  Time to improvement from 'off' to 'on'.
The duration of 'on' | 90 minutes
  The duration of 'on', the duration of time when the patient can function well.
The proportion of patients converting to 'on' any time after treatment administration. | 90 minutes
  The proportion of patients converting to 'on' any time after treatment administration.

OTHER OUTCOMES:
Safety variables | 90minutes
  Safety variables were: the pre- to post-dose change in vital signs, 12-lead ECG and continuous 12-lead Holter ECG, and lung function.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Grosset, MD, Principal Investigator — South Glasgow NHS Hospitals
Locations (9):
- Serbia (2):
  - Neurology Clinical Military Medical Academy, Crnotravska 17, Belgrade
  - Institute of Neurology Clinical Center Serbia Dr Subotica 6, Belgrade
- United Kingdom (7):
  - University Hospital, Wales, Cardiff
  - Department of Neurology, Southern General Hospital, Glasgow
  - The Walton Centre, Liverpool
  - Llandudno Hospital, Llandudno
  - Newark Hospital, Newark
  - Neurology Dept, Radcliffe Infirmary, Oxford
  - Essex Neurosciences, UnitOld Church Hospital, Essex, Romford Essex